CLINICAL TRIAL: NCT04499092
Title: COgnitive REhabilitation Treatments in Pediatric Patients with Acquired Brain Injury. from Vegetative State to Functional Recovery.
Brief Title: COgnitive REhabilitation in Pediatric Patients with ABI, from Vegetative State to Functional Recovery
Acronym: COREABI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 607rev1
Record Dates: First submitted 2020-02-25; First posted 2020-08-05 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Acquired Brain Injury; Development, Child
Keywords: Rehabilitation
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Intervention Model Description: The study will have the following steps:
  * Adaptation/preliminary validation of the CRS-R for the Italian context (typically developing children, healthy volunteers) (N=64)
  * Preliminary validation of the CRS-R in a sample of Italian patients with disorder of consciousness (N=80)
  * Evaluation and comparison of the efficacy of two multidomain neuropsychological treatments (CORE-ABI vs SET-ABI) in children emerged from a disorder of consciousness (N=40; sample size determined through power-analysis)
Who Masked: Participant, Outcomes Assessor
Masking Description: Caregivers of participants are blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Personalized neuropsychological treatment (CORE-ABI) (Active Comparator): Each patient will receive greater stimulation of the most deficient cognitive function(s), while at the same time being trained on all the other functions.
  Interventions: Other: Personalized Neuropsychological treatment (CORE-ABI)
- Sequential neuropsychological treatment (SET-ABI) (Experimental): Each patient will receive a fixed-dose stimulation of each cognitive function following a sequential order.
  Interventions: Other: Sequential Neuropsychological treatment (SET-ABI)

INTERVENTIONS:
Other: Personalized Neuropsychological treatment (CORE-ABI) — Personalized neuropsychological treatment. In the CORE-ABI intervention, the stimulation of cognitive functions will be provided based on a weekly evaluation of child's cognitive profile by a qualified neuropsychologist. Each session will have a duration of 45 min. While the first 30 minutes will be devoted to the stimulation of the most impaired cognitive function(s), the remaining 15 minutes will ensure the stimulation of the other cognitive subdomains. Domains addressed by the intervention will be the following: selective attention, sustained and divided attention, inhibition and shifting, visual-perceptual abilities, visual-spatial abilities, visual-constructional abilities, short-term memory, long-term memory, working-memory, categorization/reasoning/abstraction, problem-solving/planning and socio-emotional skills.
  Arms: Personalized neuropsychological treatment (CORE-ABI)
Other: Sequential Neuropsychological treatment (SET-ABI) — Sequential Neuropsychological Treatment. In the SET-ABI intervention, the stimulation of cognitive functions will be provided following a sequential order, identical for each child and for each session in each setting (neuropsychological treatment, speech therapy treatment and psychoeducational treatment). Each session will have a duration of 45 min.
  Specifically, the first three weeks (weeks 1-3) of treatment will target attention; in weeks 4-6, the domain of visual-spatial and visual-constructional abilities will be addressed; in weeks 7-9, memory will be the target domain; in weeks 10-12, executive functions and socio-emotional skills will be addressed.
  Arms: Sequential neuropsychological treatment (SET-ABI)

SUMMARY:
Acquired brain injuries (ABI) represent one of the most important cause of disability and mortality during the pediatric age, also in the western Countries. The important medical progress of the last decade has increased the percentages of survivals, also in patients with the most severe clinical pictures. On the other hand, a brain injury reported in the first years of life presents with a more dramatic impact on cognitive and neurological development of patients and it may significantly interfere with adjustment, vocational perspectives and quality of life. Recent studies suggest that a brain damage at an early stage of development is related to more persistent sequelae in comparison with a comparable lesion reported by an adult patient, because of the neurological immaturity of the central nervous system at the moment of the insult. Furthermore, in most cases, a brain injury is related not only to motor and sensory deficits but also to significant behavioral and cognitive problems, that may occur immediately after the acute phase and persist or worsen over the years.

DETAILED DESCRIPTION:
The aims of the present study are:

1. To contribute to the adaptation of the Italian version of the Coma Recovery Scale for pediatrics, investigating behavioral responses of children across different age and developmental levels. Typically developing children and children with disorder of cosciousness due to ABI will be included;
2. For patients with an adequate cognitive profile, to compare the efficacy of two multidomain neuropsychological interventions: a personalized neuropsychological treatment and a sequential neuropsychological treatment. In the personalized neuropsychological treatment each patient will receive greater stimulation of the most deficient cognitive function(s), while at the same time being trained on all the other functions; in the sequential neuropsychological treatment, a fixed-dose stimulation of each cognitive function following a sequential order will be provided.

ELIGIBILITY:
-For the adaptation/validation of the Coma Recovery Scale for pediatrics for the Italian context (typically developing children, healthy volunteers)

Inclusion Criteria:

* children aged between 0 and 5 years
* no suspicion of the presence of a neurodevelopmental disorder
* For the preliminary validation of the Coma Recovery Scale in clinical subjects:

Inclusion criteria:

* age between 0 and 10 years at the moment of the pathological event
* LOCFAS score <5
* a documented diagnosis of moderate-to-severe acquired brain injury of traumatic, anoxic, vascular or infective etiology (Glasgow Coma Scale, GCS<12)
* a brain lesion reported within one year from study inclusion
* For the evaluation and comparison of the efficacy of two multidomain neuropsychological treatments (CORE-ABI vs SET-ABI) in children emerged from a disorder of consciousness:
* age between 5:0 and 17:11 years at the moment of the ABI
* LOCFAS score>5
* time between ABI and assessment <3 months
* GCS <12 in the acute phase
* negative anamnesis for other developmental disorders before the ABI

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 184 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Conners Kiddie Continuous Performance Test-2nd Edition -K-CPT-2/Continuous Performance Test-3rd Edition -CPT-3 | before and immediately after the intervention
  Conners Kiddie Continuous Performance Test-2nd Edition -K-CPT-2/Continuous Performance Test-3rd Edition-CPT-3 measure sustained attention. K-CPT-2 is used with children aged up to 7:11 years, while CPT-3 is adopted with children aged 8:0-17:11 years. Scores will be expressed as T scores (M=50, SD=10). Higher scores indicate worse outcomes.

SECONDARY OUTCOMES:
BVN visual selective attention | before and immediately after the intervention
  The visual selective attention task (BVN visual selective attention) of the Italian battery 'Batteria di valutazione neuropsicologica per l'età evolutiva -BVN 5-11' [Battery for neuropsychological evaluation for developmental age -BVN 5-11] will be used for children aged 5:0-11:11 years; the same task included in the Italian battery 'Batteria di Valutazione Neuropsicologica per l'adolescenza -BVN 12-18' [Battery of neuropsychological evaluation for adolescence -BVN 12-18] will be used for children aged 12:0-17:11 years. Scores will be expressed as z-scores (M=0; SD=1), with higher scores indicating better outcomes.
Benton Judgment of Line Orientation Test | before and immediately after the intervention
  The Benton Judgment of Line Orientation Test will be used to test visual-spatial orientation. The test targets subjects from 7:0 years onwards. Scores will be expressed as z-scores (M=0; SD=1), with higher scores indicating better outcomes.
BVN Phonemic fluency | before and immediately after the intervention
  The phonemic fluency task (BVN phonemic fluency) included in the Italian 'Batteria di valutazione neuropsicologica per l'età evolutiva 5-11' [Battery for neuropsychological evaluation for developmental age -BVN 5-11] will be used for children aged 5:0-11:11 and the one included in the Italian 'Batteria di Valutazione Neuropsicologica per l'adolescenza' [Battery of neuropsychological evaluation for adolescence-BVN 12-18] will be used for children aged 12:0-17:11 years. Scores will be expressed as z-scores. (M=0; SD=1), with higher scores indicating better outcomes.
ToL Total moves | before and immediately after the intervention
  The Tower of London (ToL) will be used to assess planning and related problem-solving abilities. Total moves score will be used to evaluate the accuracy of planning. Scores will be expressed as Standard scores (M=100; SD=15) with higher scores indicating better outcomes. The administration sheet and normative data are available for children aged 7:0-15:11 years and adolescents and adults aged 16:0 years or older; thus children of this study aged less than 7:0 years will be not administered this test.
NEPSY-II Theory of Mind subscale | before and immediately after the intervention
  The 'Theory of mind' subscale of the Italian version of the battery -A Developmental NEuroPSYchological Assessment-II (NEPSY-II) will be administered. The Theory of Mind subscale-part A assesses the understanding of mental functions and other people's perspectives, with raw scores ranging from 0 to 17; the Theory of Mind subscale-part B examines the ability to match basic emotions to specific situations. Scores will be expressed as scaled scores (M=10, SD=3), ranging from 1 to 19. Higher scores indicated better outcomes. As NEPSY-II was developed and validated for children aged 3:0-16:11 years, scores of adolescents aged 17:0-17:11 years will be calculated by considering norms for adolescents aged 15:0-16:11 years.
BVN Immediate word list recall task | before and immediately after the intervention
  The BVN immediate word list recall task will be used to assess short-term verbal memory. The task included in the Italian 'Batteria di valutazione neuropsicologica per l'età evolutiva -BVN 5-11-' [Battery for neuropsychological evaluation for developmental age -BVN 5-11] will be used for children aged 5:0-11:11 years, while the one included in the Italian 'Batteria di Valutazione Neuropsicologica per l'adolescenza -BVN 12-18' ['Battery for neuropsychological evaluation for adolescence -BVN 12-18] will be used for children aged 12:0-17:11 years. Scores will be expressed as z-scores (M=0; SD=1) with higher scores indicating better outcomes.
MCST/WCST Errors | before and immediately after the intervention
  Cognitive flexibility will be assessed by using the computerized Modified Card Sorting Test (MCST) and the computerized Wisconsin Card Sorting Test (WCST). The MCST will be used for children aged 5:0-7:11, while the WCST will be used for children aged 8:0-17:11. The number of total errors (MCST/WCST errors), which represents the sum of perseverative and non-perseverative errors, will be considered for this study. Scores will be expressed as Standard scores (M=100; SD=15), with higher scores indicating better outcomes.
BVN Forward digit span | before and immediately after the intervention
  The forward digit span test will be used to assess short-term memory. The task included in the Italian 'Batteria di valutazione neuropsicologica per l'età evolutiva -BVN 5-11' [Battery for neuropsychological evaluation for developmental age -BVN 5-11] will be used for children aged 5:0-11:11 years, while the one included in the Italian 'Batteria di Valutazione Neuropsicologica per l'adolescenza -BVN 12-18' ['Battery of neuropsychological evaluation for adolescence -BVN 12-18] will be used for children aged 12:0-17:11 years. Scores will be expressed as z-scores (M=0; SD=1) with higher scores indicating better outcomes.
BVN Corsi | before and immediately after the intervention
  The Corsi block tapping task (BVN Corsi) will be used to assess visual-spatial working-memory. The task included in the Italian 'Batteria di valutazione neuropsicologica per l'età evolutiva -BVN 5-11' [Battery for neuropsychological evaluation for developmental age -BVN 5-11] will be used for children aged 5:0-11:11; the same task included in the Italian 'Batteria di Valutazione Neuropsicologica per l'adolescenza -BVN 12-18' ['Battery of neuropsychological evaluation for adolescence -BVN 12-18] will be used for children aged 12:0-17:11 years. Scores will be expressed as z-scores (M=0; SD=1) with higher scores indicating better outcomes.
Rey-Osterrieth Complex Figure Test-recall task (ROCF-recall) | before and immediately after the intervention
  The Rey-Osterrieth Complex Figure Test-recall task (ROCF-recall) will be used to evaluate long-term visual-spatial memory. In this task children will be required to reproduce a complicated line drawing 30 minutes after presentation. Scores will be expressed as z scores (M=0; SD=1), with higher scores indicating better outcomes.
Rey-Osterrieth Complex Figure Test -copy task (ROCF-copy) | before and immediately after the intervention
  The Rey-Osterrieth Complex Figure Test -copy task (ROCF-copy) will be adopted to assess visual-constructional abilities. The test targets subjects from 4:0 years onwards. Scores will be expressed as z scores (M=0; SD=1), with higher scores indicating better outcomes.
NEPSY-II Affect Recognition subscale | before and immediately after the intervention
  The 'Affect recognition' subscale of the Italian version of the battery -A Developmental NEuroPSYchological Assessment-II (NEPSY-II) will be administered. This subscale assesses the ability to recognize emotions on facial expressions. Scores will be expressed as scaled scores (M=10, SD=3), ranging from 1 to 19. Higher scores indicate better outcomes. As NEPSY-II was developed and validated for children aged 3:0-16:11 years, scores of adolescents aged 17:0-17:11 years will be calculated by considering norms for adolescents aged 15:0-16:11 years.
Test of Visual Perceptual Skills-3rd Edition -TVPS-3- | before and immediately after the intervention
  The Italian version of the Test of Visual Perceptual Skills-3rd Edition -TVPS-3- will be used to assess visual information processing. The test targets subjects from 4:0 years through 18:11. Scores will be expressed as Standard scores (M=100; SD=15), with higher scores indicating better outcomes.
ToL Initiation Time | before and immediately after the intervention
  The Tower of London (ToL) will be used to assess planning and related problem-solving abilities. Total Initiation time score will be used to evaluate the time used to planning for problem-solving. Scores will be expressed as Standard scores (M=100; SD=15) with higher scores indicating better outcomes. The administration sheet and normative data are available for children aged 7:0-15:11 years and adolescents and adults aged 16:0 years or older; thus children of this study aged less than 7:0 years will be not administered this test.
BVN Backward digit span | before and immediately after the intervention
  The Backward digit span test will be used to assess verbal working-memory. The task included in the Italian 'Batteria di valutazione neuropsicologica per l'età evolutiva -BVN 5-11' [Battery for neuropsychological evaluation for developmental age -BVN 5-11] will be used for children aged 5:0-11:11 years, while the one included in the Italian 'Batteria di Valutazione Neuropsicologica per l'adolescenza -BVN 12-18' ['Battery of neuropsychological evaluation for adolescence -BVN 12-18] will be used for children aged 12:0-17:11 years. Patients will be required to repeat a sequence of numbers presented by the examiner in a reverse order. Scores will be expressed as z-scores (M=0; SD=1) with higher scores indicating better outcomes.
BVN Delayed word list recall task | before and immediately after the intervention
  The BVN delayed word list recall task will be used to assess long-term verbal memory. The task included in the Italian 'Batteria di valutazione neuropsicologica per l'età evolutiva -BVN 5-11-' [Battery for neuropsychological evaluation for developmental age -BVN 5-11] will be used for children aged 5:0-11:11 years, while the one included in the Italian 'Batteria di Valutazione Neuropsicologica per l'adolescenza -BVN 12-18' ['Battery for neuropsychological evaluation for adolescence -BVN 12-18] will be used for children aged 12:0-17:11 years. Scores will be expressed as z-scores (M=0; SD=1) with higher scores indicating better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Eugenio Medea, Bosisio Parini, Italy, Italy

IPD SHARING:
Plan to Share IPD: No